CLINICAL TRIAL: NCT03969667
Title: Turkish Version of the Chalder Fatigue Scale: An Investigation of Its Psychometric Properties in Healthy Young Adults
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Cigdem Ayhan, associate doctor, Hacettepe University
Other Study IDs: GO 19/512
Record Dates: First submitted 2019-05-29; First posted 2019-05-31 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Fatigue; Healthy
Keywords: fatigue; assessment; reliability; validity; Chalder Fatigue Scale; Turkish version; healthy young adults
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- healthy young adults: healthy young adults

SUMMARY:
The aim of this study was to adapt the Chalder Fatigue Scale to Turkish and to examine its psychometric properties in young adults. Within the scope of the study, firstly the Turkish version of the scale will be developed and then its reliability and validity will be examined in healthy young adults in Turkey.

DETAILED DESCRIPTION:
Fatigue is a subjective experience that can affect all individuals. It is a protective symptom against physical or psychological stress for healthy individuals. However, it can negatively affect the performance of individuals in activities of daily living. In the clinic, fatigue is assessed by self-reported scales. Different fatigue scales have some advantages and disadvantages compared to each other. Moreover, it is stated that only one scale cannot fully measure the fatigue of individuals in different health status, therefore different scales have been developed.Chalder Fatigue Scale (CFS) is an easy-to-understand, short, fast and useful fatigue scale that evaluates fatigue with two dimensions (physical and mental) and enable individuals to express perceived fatigue clearly. Psychometric properties of CFS have been investigated in general population and different disease groups but not in only healthy young adults.

ELIGIBILITY:
The inclusion criteria for participants are: to be aged between 20 and 40 years old, volunteer to participate the study, able to read and speak Turkish.

Exclusion criteria are determined as individuals with known acute or chronic health conditions and illnesses and who had surgery in the past 6 months.

Further exclusion criteria are to take over-the-counter medication or food supplement, have abnormal body mass index (BMI) (lower 17 kg/m2 or higher 30 kg/m2), self reported depression as indicated by a score of > 21 on the Beck Depression Scale (BDS), pain as indicated by a score of > 0 on pain subscale of Nottingham Health Profile (NHP). Additionally, female participants were excluded if they use oral contraceptives, experience premenstrual syndrome or were pregnant within the last one year period.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community sample: The sample of the study consisted of healthy young adults, who could be announced / informed about the study and volunteered to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 353 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-02-07 (Actual)

PRIMARY OUTCOMES:
The Turkish Version of the Chalder Fatigue Scale | About 2-3 minutes
  The Chalder Fatigue Scale has a 7-item physical fatigue subscale and 4 items of mental fatigue subscale. The scale evaluates the severity of physical and mental fatigue over the last month. Each item is scored 0-3 (0=less than usual, 3=much more than usual), yielding a total between 0 and 33.
The Turkish Version of the Checklist Individual Strength Fatigue Scale | About 3-4 minutes
  The scale evaluates fatigue over the past two weeks.The questionnaire consists of 20 items with a 7-point Likert scale scoring. A total score is derived by summation of the item scores (20-140). There are four subscales; Fatigue Severity, measuring the subjective experience of fatigue (8 items); Concentration, measuring concentration problems (5 items); Motivation, measuring reduced motivation (4 items) and Activity, measuring the reduction of activities (3 items).

SECONDARY OUTCOMES:
Visual Analog Scale to Evaluate Physical and Mental Fatigue | About 1 minutes
  Self reported physical and mental fatigue severity over the last month. It is scored 0=no fatigue; 10= tired as bad as can be
The Turkish Version of the Pittsburgh Sleep Quality Index | About 2-3 minutes
  The scale assesses sleep quality over a 1-month period. The questionnaire consists of 19 self-rated questions and 5 questions that should be answered by roommates. The latter questions are used only for clinical information. The 19 questions are categorized into 7 components, graded on a score that ranges from 0 to 3. The scale's components are as follows: subjective sleep quality (C1), sleep latency (C2), sleep duration (C3), habitual sleep efficiency (C4), sleep disturbances (C5), use of sleeping medication (C6) and daytime dysfunction (C7). The sum of scores for these 7 components yields one global score, which ranges from 0 to 21, where the highest score indicates worst sleep quality.
The Turkish Version of the Beck Depression Inventory | About 4-5 minutes
  It is a 21-item self-report questionnaire for assessing the severity of depressive symptoms over past week; the items comprise four ordinal categories (from 0 through 3). Absence (or "as usual") of depressive symptom in each item is scored as "0" and presence of symptom is scored between 1 and 3, with the higher score indicating more intense symptom severity. The possible total score ranges from 0 to 63.
The Turkish Version of the Nottingham Health Profile | About 4-5 minutes
  The scale measures subjective health status using 38 items that assess 6 subscales (physical mobility, pain, energy level, sleep, emotional reaction and social isolation); each question answered by (yes) or (no) with each question assigned a weighted value. Scores for each section can range from 0 "no problems" to 100 "all problems listed are present" where the sum of all weighted values in a given subscale adds up to 100.

CONTACTS AND LOCATIONS:
Overall Officials: Cigdem Ayhan, Assoc. Prof., Principal Investigator — Hacettepe University; Ridvan M Adin, R. A., Study Chair — Hacettepe University; Ali N Ceren, R. A., Study Chair — Hacettepe University; Ayla Fil Balkan, Asst. Prof., Study Chair — Hacettepe University; Yeliz Salci, Asst. Prof., Study Chair — Hacettepe University; Kadriye Armutlu, Prof., Study Chair — Hacettepe University
Locations (1):
- Hacettepe University Faculty of Health Sciences Department of Physiotherapy and Rehabilitation, Ankara, Altındag, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mota DD, Pimenta CA. Self-report instruments for fatigue assessment: a systematic review. Res Theory Nurs Pract. 2006 Spring;20(1):49-78. doi: 10.1891/rtnp.20.1.49. PMID 16544894
- [Background] Beydoun J, Nasrallah L, Sabrah T, Caboral-Stevens M. Towards a Definition of Caregiver Fatigue: A Concept Analysis. ANS Adv Nurs Sci. 2019 Oct/Dec;42(4):297-306. doi: 10.1097/ANS.0000000000000262. PMID 30839335
- [Background] Glaus A, Crow R, Hammond S. A qualitative study to explore the concept of fatigue/tiredness in cancer patients and in healthy individuals. Eur J Cancer Care (Engl). 1996 Jun;5(2 Suppl):8-23. doi: 10.1111/j.1365-2354.1996.tb00247.x. PMID 9117043
- [Background] Engberg I, Segerstedt J, Waller G, Wennberg P, Eliasson M. Fatigue in the general population- associations to age, sex, socioeconomic status, physical activity, sitting time and self-rated health: the northern Sweden MONICA study 2014. BMC Public Health. 2017 Aug 14;17(1):654. doi: 10.1186/s12889-017-4623-y. PMID 28806984
- [Background] Cella M, Chalder T. Measuring fatigue in clinical and community settings. J Psychosom Res. 2010 Jul;69(1):17-22. doi: 10.1016/j.jpsychores.2009.10.007. Epub 2009 Dec 11. PMID 20630259
- [Background] Zwarts MJ, Bleijenberg G, van Engelen BG. Clinical neurophysiology of fatigue. Clin Neurophysiol. 2008 Jan;119(1):2-10. doi: 10.1016/j.clinph.2007.09.126. Epub 2007 Nov 26. PMID 18039594
- [Background] Chalder T, Berelowitz G, Pawlikowska T, Watts L, Wessely S, Wright D, Wallace EP. Development of a fatigue scale. J Psychosom Res. 1993;37(2):147-53. doi: 10.1016/0022-3999(93)90081-p. PMID 8463991
- [Background] Beaton DE, Bombardier C, Guillemin F, Ferraz MB. Guidelines for the process of cross-cultural adaptation of self-report measures. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3186-91. doi: 10.1097/00007632-200012150-00014. No abstract available. PMID 11124735
- [Background] Dittner AJ, Wessely SC, Brown RG. The assessment of fatigue: a practical guide for clinicians and researchers. J Psychosom Res. 2004 Feb;56(2):157-70. doi: 10.1016/S0022-3999(03)00371-4. PMID 15016573
- [Background] Ergin G, Yildirim Y. A validity and reliability study of the Turkish Checklist Individual Strength (CIS) questionnaire in musculoskeletal physical therapy patients. Physiother Theory Pract. 2012 Nov;28(8):624-32. doi: 10.3109/09593985.2011.654321. Epub 2012 Feb 10. PMID 22324761
- [Background] Kucukdeveci AA, McKenna SP, Kutlay S, Gursel Y, Whalley D, Arasil T. The development and psychometric assessment of the Turkish version of the Nottingham Health Profile. Int J Rehabil Res. 2000 Mar;23(1):31-8. doi: 10.1097/00004356-200023010-00004. PMID 10826123
- [Background] Wood C, Magnello ME, Jewell T. Measuring vitality. J R Soc Med. 1990 Aug;83(8):486-9. doi: 10.1177/014107689008300803. PMID 2231574

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-21): https://cdn.clinicaltrials.gov/large-docs/67/NCT03969667/Prot_SAP_001.pdf